CLINICAL TRIAL: NCT02617238
Title: Strategy for Preventing Cardiovascular and Renal Events Based on ARTErial Stiffness
Acronym: SPARTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); Fondation pour la Recherche en Hypertension Artérielle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K110102
Record Dates: First submitted 2015-09-15; First posted 2015-11-30 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: arterial stiffness; cardiovascular risk; cardiovascular events; renal events
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PWV group (Active Comparator): Cardiovascular risk management based on PWV will include altogether
  1. the implementation of international guidelines,
  2. the normalisation of blood pressure, and
  3. the normalisation of arterial stiffness
  Interventions: Other: Cardiovascular risk management based on PWV
- Conventional group (No Intervention): These patients will be treated according to the 2007 (and then 2013) ESH-ESC Guidelines for the management of hypertension

INTERVENTIONS:
Other: Cardiovascular risk management based on PWV — Arterial stiffness will be measured through the determination of the carotid-femoral pulse wave velocity (PWV).
  1. In the "PWV group", PWV will be measured at baseline, and then every 6 months. PWV measurement will guide the intensification of treatment. Measurements will be immediately available to the physician in charge of the patient, in order to adapt treatment. The therapeutic strategy is based both on the normalisation of BP and then on the BP-independent reduction in PWV, using commercially available antihypertensive medications.
  2. In the "conventional group", PWV will be measured at baseline, after 2 years, and at the end of the study. PWV values will be masked to the physician
  Arms: PWV group

SUMMARY:
Randomised two parallel groups multicenter study using a Prospective Randomised Open Blinded End-point design (PROBE), aiming at comparing the efficacy of a therapeutic strategy targeting the normalisation of arterial stiffness for reducing cardiovascular (CV) and renal events, in comparison with a classical therapeutic strategy implementing the European Society of Hypertension-European Society of Cardiology (ESH-ESC) Guidelines, in patients with essential hypertension and medium-to-very high CV risk.

DETAILED DESCRIPTION:
The objective is to show that a therapeutic strategy targeting the implementation of international guidelines PLUS the normalisation of blood pression (BP < 140 and 90 mmHg) plus the normalisation of arterial stiffness (measured every 6 months) Pulse Wave Velocity group (PWV group) reduces CV and renal events to a significantly greater extent than the sole implementation of Guidelines (conventional group, with PWV measurement at baseline and every 2 years).

Experimental design: Prospective Randomised Open Blinded Endpoint (PROBE) multicenter, two parallel groups, study.

Therapeutic strategy in the PWV group:

1. Use maximal recommended doses of angiotensin-converting-enzyme inhibitor (ACEIs) or Angiotensin II receptor blockers (ARBs) as first step treatment. And then adapt treatment to PWV values.
2. In second step, use combination therapy with Calcium channel blockers (CCBs)
3. Use diuretics in combination therapy, either as an alternative to CCBs in second step or as triple therapy in third step
4. Use, as fourth step, vasodilating beta-blockers (VD-BB) or spironolactone
5. In parallel, correct all CV risk factors according to ESH-ESC Guidelines, and reinforce treatment (hypolipidemic drugs, glucose lowering drugs, antiplatelets) if secondary prevention.

Therapeutic strategy in the conventional group: Apply the ESH-ESC Guidelines

ELIGIBILITY:
Inclusion Criteria:

* registration to the French social security system
* patients who did not specifically express their non willingness to participate

PLUS either A, B or C:

1. Patients with essential hypertension, aged 55 to 75 years old, both sexes

   * Grade 1 hypertension of more
   * Treated or not
   * Whatever the control of BP
   * Under primary of secondary prevention (more than 3 months stroke or myocard infarctus (MI), or stable angina or peripheral artery disease) PLUS at least 3 CV risk factors according to ESH-ESC 2007 guidelines or metabolic syndrome associating at least 2 of the following criteria

     * SBP/DBP over 130/85 mmHg
     * HDL-C <1.0 mmol/l (0,4 g/l) (M) or < 1.2 mmol/l (0,46 g/l) (F)
     * Triglycerides >1,7 mmol/l (>1,5 g/l)
     * Fasting blood glucose 5,6 - 6,9 mmol/l (1,02-1,25 g/l)
     * Waist circumference > 102 cm (M) ou 88 cm (F) or Type 2 diabetes or Target organ damage, according to the definition of the ESH-ESC Guidelines for the Management of Hypertension or CV disease or chronic kidney disease
2. SBP > 180 mmHg and/or DBP > 110 mmHg
3. SBP > 160 mmHg AND DBP < 70 mmHg

Exclusion Criteria:

* Patients with ABPM or self-measurement normal without treatment (<130 mmHg and 80 in the ABPM 24 or <135 and 85 mmHg or daytime ABPM self-measurement of blood pressure)
* Patients with secondary hypertension (renal artery stenosis, pheochromocytoma, or hypermineralocortisism)
* Patients with hypertension secondary to diabetic nephropathy
* Patients aged under 55 or over 75 years,
* Low-risk CV patients
* Patients with severe chronic renal impairment creatinine clearance (MDRD) <30ml / min / 1.73m2
* Patients with type I diabetes
* Patients with severe disease threatening the vital prognosis in the short and medium terms
* Patients who previously experienced a painful gynecomastia under spironolactone
* Patients with alcohol dependence or excessive consumption alcoholic beverages (at the judgement of the investigator)
* patients with accident history neurovascular, coronary insufficiency (coronary bypass surgery or percutaneous coronary intervention) not older than 3 month
* Patients with a history of acute heart failure or having open failure heart (NYHA class III-IV)
* Patients with unstable angina
* Auricular Fibrillation (AF) less than 6 months ago
* Patients with aortic stent
* Patients with known aneurysms of the abdominal aorta
* Patients with atrioventricular block second or third degree without pacemaker
* Patients having received organ transplant or placed on a waiting list for transplantation
* Patients with severe chronic inflammatory disease (rheumatoid arthritis; lupus; scleroderma ...)
* Patients with severe chronic infectious disease
* Patients who have had an MI less than 3 months ago
* Patients with stroke there are less than 3 months ago
* Patients with progression of peripheral arterial disease
* Patient whose pregnancy is known or which has no effective contraception if is of childbearing age, or if she is breastfeeding
* Patients who have expressed their opposition to participate in the protocol or have an inability to understand or follow the protocol
* The patients geographically too far from the place of investigation
* Patients already participating in other drug research protocol or Interventional

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of cardiovascular and renal events | 4 years of follow-up
  The primary efficacy outcome variable is defined as the composite endpoint of cardiovascular death, non-fatal myocardial Infarction, non-fatal stroke, adverse renal outcome (defined by chronic dialysis, kidney transplantation, or doubling of serum creatinine) and hospitalization for any of the following causes: angioplasty or bypass surgery for coronary or peripheral vessel disease, congestive heart failure, or aortic dissection. An independent committee will validate the events and causes blinded treatment received

SECONDARY OUTCOMES:
Number of non-fatal myocardial Infarction | 4 years follow-up
Number of non-fatal stroke | 4 years follow-up
Number of adverse renal outcome (defined by chronic dialysis, kidney transplantation, or doubling of serum creatinine) | 4 years follow-up
Number of hospitalization for any of the following causes: angioplasty or bypass surgery for coronary or peripheral vessel disease | 4 years follow-up
Number of congestive heart failure | 4 years follow-up
Number of aortic dissection | 4 years follow-up
Carotid-femoral pulse wave velocity (PWV) value at the end of the study | 4 years follow-up
Central systolic blood pressure value | 4 years follow-up
Central pulse pressure value | 4 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LAURENT, MD, PhD, Principal Investigator — Hopital Europen Georges Pompidou, Assistance publique Hopitaux de Paris; Pierre BOUTOUYRIE, MD, PhD, Study Director — Hopital Europen Georges Pompidou, Assistance publique Hopitaux de Paris
Locations (1):
- Clinical Investigation Center, Hopital Europeen Georges Pompidou, Paris, France

REFERENCES:
- [Background] Laurent S, Briet M, Boutouyrie P. Arterial stiffness as surrogate end point: needed clinical trials. Hypertension. 2012 Aug;60(2):518-22. doi: 10.1161/HYPERTENSIONAHA.112.194456. Epub 2012 Jun 25. No abstract available. PMID 22733473
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527